CLINICAL TRIAL: NCT03245437
Title: Effects of Oxytocin on Social Cognition Training: Relationship to Target Engagement
Brief Title: Target Engagement and Response to Oxytocin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen R. Marder, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT R33; R33MH107564 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: Social Cognition; Oxytocin
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oxytocin with SCST (Experimental): Oxytocin with SCST (active condition)
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Social Cognition Skills Training
- Oxytocin with Health Management (Sham Comparator): Administration of OT with control psychosocial treatment
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Health Management
- Placebo with SCST (Placebo Comparator): Administration of Placebo with active psychosocial treatment
  Interventions: Behavioral: Social Cognition Skills Training; Drug: Placebo nasal spray
- Placebo with HM (Placebo Comparator): Administration of Placebo with control psychosocial treatment
  Interventions: Behavioral: Health Management; Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — nasal spray
  Other Names: OT
  Arms: Oxytocin with Health Management; Oxytocin with SCST
Behavioral: Social Cognition Skills Training — Group based training in social cognition skills
  Other Names: SCST
  Arms: Oxytocin with SCST; Placebo with SCST
Behavioral: Health Management — Group-based training in mental health management
  Other Names: HM
  Arms: Oxytocin with Health Management; Placebo with HM
Drug: Placebo nasal spray — placebo condition
  Other Names: PBO
  Arms: Placebo with HM; Placebo with SCST

SUMMARY:
This study will measure whether the engagement of intranasal oxytocin with a brain target is related to effects on learning during a social cognition training program.

DETAILED DESCRIPTION:
The study will determine whether oxytocin (OT) administration 30 min before a training session enhances the learning of social information in the context of a social cognitive skills training (SCST) program, and it will test a possible mediator of this effect. Subjects with psychotic disorders will be randomized to one of four groups in a 2 by 2 factorial design: OT with SCST; Placebo with SCST; OT with training control condition; placebo with training control condition. Target engagement will be measured in an OT challenge (placebo versus OT one week apart) prior to baseline assessment. The measure of target engagement will be EEG mu suppression while observing biological motion. A social cognition battery will be administered at baseline, at midpoint after 6 weeks of SCST, and at completion of training at 12 weeks. The battery will include measures of social cue identification and mentalizing.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder
* stable on an antipsychotic medication

Exclusion Criteria:

* positive pregnancy test history of head injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Social Cognition Composite Score | 16 weeks
  We will assess social cognition in two subdomains: (1) social cue identification (Managing Emotions component of Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) branch 1, Ekman, Profile of Nonverbal Sensitivity (PONS); and (2) mentalizing (The Awareness of Social Inference Test (TASIT). and Empathic accuracy) (see below). The primary summary measure for each test will be mean-centered and standardized to create a Z-score. These Z-scores will be averaged to create a single composite score for social cognition that will serve as the primary outcome measure.

SECONDARY OUTCOMES:
Composite score of non-social cognition from the MATRICS Consensus Cognitive Battery | 16 weeks
  Standardized z-score

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Marder, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States